CLINICAL TRIAL: NCT01403259
Title: Phase II Study of SOX in Patients With Platinum-resistant Nasopharyngeal Carcinoma
Brief Title: SOX as Salvage Treatment in Nasopharyngeal Carcinoma
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: poor accrual of eligible patients
Sponsor: Fudan University (Other)
Responsible Party: Principal Investigator, Ye Guo, Dr., Fudan University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HNTG 11-02
Record Dates: First submitted 2011-07-26; First posted 2011-07-27 (Estimated); Last update posted 2014-08-20 (Estimated); Status verified 2014-08

CONDITIONS: Nasopharyngeal Carcinoma
Keywords: Nasopharyngeal carcinoma; S-1; Oxaliplatin
MeSH Terms: conditions — Nasopharyngeal Carcinoma | interventions — S 1 (combination); Oxaliplatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- S-1 plus oxaliplatin (Experimental): S-1 60 mg BID at day 1-14 Oxaliplatin 100 mg/m2 at day 1 Frequence of cycles: every 3 weeks for 6 cycles
  Interventions: Drug: S-1 plus oxaliplatin

INTERVENTIONS:
Drug: S-1 plus oxaliplatin — S-1 60 mg BID at day 1-14 Oxaliplatin 100 mg/m2 at day 1 Frequence of cycles: every 3 weeks
  Other Names: S-1; Oxaliplatin

SUMMARY:
The aim of the study is to evaluate the efficacy and safety of SOX regimen (S-1 plus oxaliplatin) as salvage treatment in patients with relapsed or metastatic nasopharyngeal carcinoma.

DETAILED DESCRIPTION:
The treatment option in patients with platinum-resistant relapsed or metastatic nasopharyngeal carcinoma is limited. Previous studies showed that both S-1 and oxaliplatin were effective in head and neck cancer. Moreover, SOX (S-1 plus oxaliplatin) was proved to be tolerable in advanced stage gastric cancer. Therefore, we aim to evaluate this regimen in salvage setting of nasopharyngeal carcinoma.

ELIGIBILITY:
Inclusion Criteria:

* Age range: 18-75 years old
* Histological confirmed incurable relapsed or metastatic nasopharyngeal carcinoma
* Prior exposure of at least one line of platinum-containing regimen
* ECOG performance status 0-1
* Life expectancy of more than 3 months
* Bone marrow function: ANC≧1.5×109/L, PLT≧100×109/L, Hb≧80g/L
* Liver function: total bilirubin, ALT and AST <1.5×UNL
* Renal function: Cr<1.5×UNL, CCR≧50ml/min
* Without > 1 grade of neuropathy

Exclusion Criteria:

* With curable treatment option
* With CNS involvement
* Prior platinum exposure only in neo-adjuvant/adjuvant setting or concurrently used with radiotherapy
* Treated with > 2 lines of palliative chemotherapy
* With prior exposure of S-1 or oxaliplatin
* History of other malignancies except cured basal cell carcinoma of skin and carcinoma in-situ of uterine cervix
* Significant active infection
* Pregnant or lactating women

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2011-07; Primary Completion 2014-12 (Estimated); Study Completion 2015-12 (Estimated)

PRIMARY OUTCOMES:
Median progression-free survival | 1 year

SECONDARY OUTCOMES:
Overall response rate | 6 weeks
Median overall survival | 1.5 year

CONTACTS AND LOCATIONS:
Overall Officials: Ye Guo, MD, Principal Investigator — Fudan University
Locations (1):
- Fudan University Shanghai Cancer Center, Shanghai, China